CLINICAL TRIAL: NCT01394640
Title: Evaluation of Immunologic Response After Pandemic Influenza A (H1N1) Vaccine in Oncologic and Hematologic Patients
Brief Title: Immunologic Response After Pandemic Influenza A (H1N1) Vaccine in Onco- Hematologic Patients
Status: Completed | Type: Observational
Sponsor: Paolo Corradini (Other)
Responsible Party: Sponsor-Investigator, Paolo Corradini, Professor, Fondazione IRCCS Istituto Nazionale dei Tumori, Milano
Organization: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Other Study IDs: INT 72/09
Record Dates: First submitted 2011-07-11; First posted 2011-07-14 (Estimated); Last update posted 2024-01-09 (Actual); Status verified 2024-01

CONDITIONS: Lymphoma; Multiple Myeloma; Myeloproliferative Disease
MeSH Terms: conditions — Lymphoma; Multiple Myeloma; Myeloproliferative Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum and blood sample
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Healthy Volunteers: Healthy people without any serious comorbidity (no immunosuppressive treatment, no autoimmune disease, no cancer) receiving the same vaccine
  Interventions: Biological: Reassortant vaccine virus NYMC X-179A (New York Medical College, New York) derived form the A/california/7/2009 (H1N1) virus
- Onco-hematologic patients: Patients with lymphoma or myeloproliferative diseases or multiple myeloma either receiving chemotherapy or in follow-up or treated with allogeneic hematopoietic stem cell transplant.
  Interventions: Biological: Reassortant vaccine virus NYMC X-179A (New York Medical College, New York) derived form the A/california/7/2009 (H1N1) virus

INTERVENTIONS:
Biological: Reassortant vaccine virus NYMC X-179A (New York Medical College, New York) derived form the A/california/7/2009 (H1N1) virus — The vaccine was administered intramuscularly as a single dose of 7.5 ug of hemagglutinin antigen.
  Other Names: Vaccine against A/H1N1 influenza

SUMMARY:
Primary objective

1) To assess whether oncologic and hematologic patients develop a protective immunological response after pandemic Influenza A (H1N1) vaccine

Secondary objectives

1. To compare the levels of antibody response against A (H1N1) influenza virus between oncologic and hematologic patients relative to a cohort of healthy volunteers
2. To assess the incidence of A (H1N1) infection in vaccinated oncologic and hematologic patients in comparison with a cohort of vaccinated healthy volunteers. To assess the clinical symptoms attributable to influenza infection in vaccinated oncologic and hematological patients and healthy volunteers.
3. To compare the levels of antibody response against A (H1N1) influenza virus between the following subgroups: patients with ongoing chemotherapy; patients who have completed the chemotherapy treatment; patients treated with autologous or allogeneic peripheral blood hematopoietic stem cell transplant (PBSCT)

Study procedures: Onco-hematological patients will perform a blood sample collection before the vaccination, on day +21 after vaccination , on day +50 and on day +90. At the end of the collection, the investigators will perform immunological test to evaluate the antibody titer and the cellular response. The titer of antibodies against the vaccine strain will be measured in all samples by hemagglutination-inhibition (HI) assays with the use of turkey erythrocytes and according to EMEA guidelines. Response criteria will be the achievement of a protective title of HI test > 1:40. In addition, the investigators will evaluate: geometric mean titers and a fourfold titer increase compared with prevaccination titers. Cellular-mediated response will be analysed by flow-cytometry. A control cohort of healthy volunteers who received A(H1N1) vaccine will perform the same blood sample collection.

Evaluation of clinical response: Oncologic and hematologic patients will be followed as outpatients or inpatients according to routine controls for their disease. In case that symptoms of the upper airways or influenza-like symptoms develop, the symptoms will be recorded in the clinical database, nasal and pharyngeal swaps will be performed according to the doctor who is taking care of the patient. In order to evaluate the clinical efficacy of the vaccination, the swaps will be tested for A (H1N1) influenza virus infection. No further studies will be performed after 3 months from the vaccination.

DETAILED DESCRIPTION:
Primary objective

1) To assess whether oncologic and hematologic patients develop a protective immunological response after pandemic Influenza A (H1N1) vaccine Secondary objectives

1. To compare the levels of antibody response against A (H1N1) influenza virus between oncologic and hematologic patients relative to a cohort of healthy volunteers
2. To assess the incidence of A (H1N1) infection in vaccinated oncologic and hematologic patients in comparison with a cohort of vaccinated healthy volunteers. To assess the clinical symptoms attributable to influenza infection in vaccinated oncologic and hematological patients and healthy volunteers.
3. To compare the levels of antibody response against A (H1N1) influenza virus between the following subgroups: patients with ongoing chemotherapy; patients who have completed the chemotherapy treatment; patients treated with autologous or allogeneic peripheral blood hematopoietic stem cell transplant (PBSCT) Study population and design

The study population consists consecutive patients with oncologic or hematologic diseases who are planned to receive A (H1N1) influenza vaccine

Study procedures The patients will perform a blood sample collection (serum vial) on day 0 (range: 0- 2 days before vaccination) before the vaccination, a blood sample collection (serum vial) on day +21 (range: +/- 5 days) after vaccination , a blood sample collection (serum vial) on day +50 (range: +/- 5 days) and on day +90 range: +/- 5 days) after vaccination. The samples will be frozen in 500 mcl aliquots at -20°C. At the end of the collection we will perform immunological test to evaluate the antibody titer and the cellular response. The serum samples will be stored at the laboratory of Virology of the University of Milan. The titer of antibodies against the vaccine strain will be measured in all samples by means of hemagglutination-inhibition (HI) assays with the use of turkey erythrocytes and according to EMEA guidelines. Response criteria will be the achievement of a protective title of HI test > 1:40. In addition we will evaluate: geometric mean titers and a fourfold titer increase compared with prevaccination titers. Cellular-mediated response will be analysed by incubating CD3+ patients' cells with influenza A Antigens and evaluation of: 1) cellular expansion by flow-cytometry analysis of dilution of carboxyfluorescein succinimidyl ester (CFSE); 2) IFN-gamma production by ELISPOT.

A control cohort of healthy volunteers who received A(H1N1) vaccine will perform the same blood sample collection in order to compare the immunological response between oncologic and hematologic patients relative to healthy cohort.

Evaluation of clinical response:

Oncologic and hematologic patients will be followed as outpatients or inpatients according to routine controls for their disease. In case that symptoms of the upper airways or influenza-like symptoms develop, the symptoms will be recorded in the clinical database, nasal and pharyngeal swaps will be performed according to the doctor who is taking care of the patient. In order to evaluate the clinical efficacy of the vaccination, the swaps will be tested for A (H1N1) influenza virus infection.

No further studies will be performed after 3 months from the vaccination.

Sample size The trial will accrue 25 patients for each subpopulation to be analyzed. This sample size has a 90% power to evaluate an increase of the probability to have a biological response from a theoretical value of 20% (low efficacy of the vaccine) to a value of 50% (target of effectiveness) at the 5% significance (student t test, one tail). The subpopulations are as follows: patients with ongoing chemotherapy; patients who have completed the chemotherapy treatment; patients treated with autologous or allogeneic transplant of hematopoietic stem cell.

We will accrue a "calibration" group comprising at least 100 healthy volunteers. This group will comprise people working at the National Cancer Institute in Milan who have signed an informed consent to participate to the study. This size of the sample allows a precision on the evaluation of the probability of obtaining a biological response (half of the confidence interval) that is not lower than 10%

Study duration The estimated duration of enrolment is of 6 months. The enrolment of the hematologic and oncologic patients and of the cohort of healthy volunteers will be performed in 3 months and the study will be closed on day +90 with a blood sample collection.

Selection criteria Inclusion criteria

* Age ≥18 years
* Oncologic and hematologic patient with the plan of receiving the A (H1N1) vaccine
* Control Group: a silent history for oncologic and hematologic diseases; planned of receiving the A (H1N1) vaccine
* Written informed consent

Exclusion criteria

* Infusion of human Immunoglobulin ongoing or within prior 30 days
* Therapy with monoclonal or polyclonal antibodies ongoing or within prior 30 days
* Therapy with IL-1 or IL-2 or IFN-gamma ongoing or within prior 30 days
* Autologous PBSCT less than 1 month or Allogeneic PBSCT less than 6 months
* Pregnancy or lactation
* Type I hypersensitivity
* Ongoing Anticoagulant therapy or platelets < 50000/ul

Study Procedures at baseline: Medical history for oncologic and hematologic disease; gynecologic history for women under 50 years of age

• Serum sample on the day of vaccination or 2 days in advance

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Oncologic and hematologic patient with the plan of receiving the A (H1N1) vaccine
* Control Group: a silent history for oncologic and hematologic diseases; planned of receiving the A (H1N1) vaccine
* Written informed consent

Exclusion Criteria:

* Infusion of human Immunoglobulin ongoing or within prior 30 days
* Therapy with monoclonal or polyclonal antibodies ongoing or within prior 30 days
* Therapy with IL-1 or IL-2 or IFN-gamma ongoing or within prior 30 days
* Autologous PBSCT less than 1 month or Allogeneic PBSCT less than 6 months
* Pregnancy or lactation
* Type I hypersensitivity
* Ongoing Anticoagulant therapy or platelets < 50000/ul

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy, nonpregnant adults, or patients affected by hematologic malignancies and older than 18 years, were eligible.
Sampling Method: Non-Probability Sample
Enrollment: 124 (Actual)
Dates: Start 2009-10; Primary Completion 2010-05 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
To assess antibody response (antibody titer > 1:40 or four-fold increase, geometric mean titer) in onco-hematologic patients and controls and whether this response changes over time | Day 0, 30, 60, 90
  The antibody titers against virus A/H1N1 will be measured in all samples by means of hemagglutination-inhibition (HI) assays with the use of turkey erythrocytes and according to EMEA guidelines. Antibody titers in control, patients and in different patient subgroups will be compared on different time points.

SECONDARY OUTCOMES:
To assess virus specific cell mediated response (by flow-cytometry evaluation) in onco-hematologic patients and controls and whether this response changes over time. | 0, 30, 60, 90
  Cellular-mediated response will be analysed by incubating CD3+ cells with influenza A Antigens and evaluation of: 1) cellular expansion by flow-cytometry analysis of dilution of carboxyfluorescein succinimidyl ester (CFSE); 2) IFN-gamma production by ELISPOT.
To assess whether controls or patients develop influenza like illness or symptoms. | Day 0, 30, 60, 90
  Subjects will be required to report the occurrence of symptoms suggestive for an influenza-like illness. An influenza-like illness is defined as an oral temperature of more than 38°C or a history of fever or chills and at least one influenza-like symptom.
  In case of symptoms of the upper airways or influenza-like symptoms, nasal and pharyngeal swaps will be performed and tested for A (H1N1) influenza virus infection.

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Corradini, MD, Principal Investigator — Fondazione IRCCS Istituto Nazionale dei Tumori, Milano
Locations (1):
- Fondazione IRCCS Istituto Nazionale dei Tumori, Milan, Italy

REFERENCES:
- [Background] Kunisaki KM, Janoff EN. Influenza in immunosuppressed populations: a review of infection frequency, morbidity, mortality, and vaccine responses. Lancet Infect Dis. 2009 Aug;9(8):493-504. doi: 10.1016/S1473-3099(09)70175-6. PMID 19628174
- [Background] Zhu FC, Wang H, Fang HH, Yang JG, Lin XJ, Liang XF, Zhang XF, Pan HX, Meng FY, Hu YM, Liu WD, Li CG, Li W, Zhang X, Hu JM, Peng WB, Yang BP, Xi P, Wang HQ, Zheng JS. A novel influenza A (H1N1) vaccine in various age groups. N Engl J Med. 2009 Dec 17;361(25):2414-23. doi: 10.1056/NEJMoa0908535. Epub 2009 Oct 21. PMID 19846844
- [Background] Greenberg ME, Lai MH, Hartel GF, Wichems CH, Gittleson C, Bennet J, Dawson G, Hu W, Leggio C, Washington D, Basser RL. Response to a monovalent 2009 influenza A (H1N1) vaccine. N Engl J Med. 2009 Dec 17;361(25):2405-13. doi: 10.1056/NEJMoa0907413. Epub 2009 Sep 10. PMID 19745216